CLINICAL TRIAL: NCT07352943
Title: Development of a Mindfulness-Based Smartphone Application for BMT Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23529
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Caregivers of Hematopoietic Stem Cell Transplant (HCT) Patients
MeSH Terms: interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App (Experimental): Participants receive access to the smartphone application, a 6-week mindfulness-based behavioral intervention adapted from the FOCUS program. Caregivers begin using the app the week prior to the patient's hematopoietic stem cell transplant and continue through six weeks of daily modules that include audio meditations, videos, text-based content, and reflection exercises.
  Interventions: Behavioral: App

INTERVENTIONS:
Behavioral: App — A smartphone-delivered mindfulness program providing daily modules, guided meditations, brief strategies, and reflection prompts designed to reduce caregiver burden and distress.

SUMMARY:
This pilot study evaluates the feasibility, acceptability, usability, and engagement of a smartphone-delivered mindfulness intervention for caregivers of hematopoietic stem cell transplant (HCT) patients. Thirty caregivers will use the app for six weeks beginning the week prior to the patient's transplant. Participants will complete baseline and end-of-treatment surveys and a brief qualitative interview.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Identified caregiver of a patient scheduled for HCT at Moffitt Cancer Center
* Able to provide informed consent
* Able to read and write in English
* Owns a smartphone and willing to download the study app

Exclusion Criteria:

* None beyond failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | During the enrollment period (anticipated 6-8 months)
  Recruitment will be assessed by the ability to recruit approximately 4 caregivers per month until the target sample of 30 is reached.
Feasibility: Retention Rate | Baseline to 6 weeks
  Percentage of enrolled participants who complete the study through the end-of-treatment.
Feasibility: Survey Completion | Baseline and 6 weeks
  Percentage of participants who complete the baseline REDCap survey and the end-of-treatment survey.
Acceptability: System Usability Scale (SUS) | 6 weeks
  Usability of the app measured using the System Usability Scale.
Engagement: Module Completion Rate | 6 weeks
  Number of modules completed per week.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided